CLINICAL TRIAL: NCT02499107
Title: The Effects of Potatoes and Other Carbohydrate Side Dishes Consumed With Meat on Food Intake, Glycaemia and Satiety Response in Children
Brief Title: The Effects of Carbohydrate Source on Food Intake, Blood Glucose and Gut Hormone Response in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: APRE_29695
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Diabetes
Keywords: food intake; satiety; blood glucose; potato; insulin
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Rice treatment (Experimental): Dietary Intervention: Ad libitum intake of white rice
  Interventions: Dietary Supplement: Rice treatment
- Pasta treatment (Experimental): Dietary Intervention: Ad libitum intake of pasta
  Interventions: Dietary Supplement: Pasta treatment
- boiled and mashed potato treatment (Experimental): Dietary Intervention: Ad libitum intake of boiled and mashed potato
  Interventions: Dietary Supplement: Boiled and mashed potato treatment
- Baked french fries treatment (Experimental): Dietary Intervention: Ad libitum intake of baked french fries
  Interventions: Dietary Supplement: Baked french fries treatment
- Fried french fries treatment (Experimental): Dietary Intervention: Ad libitum intake of fried french fries
  Interventions: Dietary Supplement: Fried french fries treatment

INTERVENTIONS:
Dietary Supplement: Rice treatment — All arms are given to all participants, in a randomized (cross over) order
  Arms: Rice treatment
Dietary Supplement: Pasta treatment
  Arms: Pasta treatment
Dietary Supplement: Boiled and mashed potato treatment
  Arms: boiled and mashed potato treatment
Dietary Supplement: Baked french fries treatment
  Arms: Baked french fries treatment
Dietary Supplement: Fried french fries treatment
  Arms: Fried french fries treatment

SUMMARY:
This study will compare the effects of commonly consumed carbohydrate sources such as potatoes, pasta and rice along with a fixed portion of meat on blood glucose, satiety and insulin levels among healthy body weight children. Healthy boys and girls, aged between 11 - 13 years old, will be involved in this study.

DETAILED DESCRIPTION:
The prevalence of childhood obesity and overweight has become a major health concern worldwide. Prevention of overweight and obesity in children is a high priority because they are at high risk of becoming obese adults and obesity is predictive of the development of coronary heart disease, hypertension and diabetes. Thus, there is a need for food-based solutions to increase satiety and subsequently reduce energy intake.

Over the past 40 years, the consumption of potatoes has decreased by 41% which may be a consequence of movements aimed at decreasing serving sizes, or the outright banning, of potato foods from cafeterias and quick service restaurants such as French fries due to the observational studies showing they are linked with increased risk of obesity. Alternate energy dense starches such as rice and pasta have increased in consumption as a result for meal accompaniments with no discernible decrease in the upward trajectory of the number of overweight and obese individuals. These recent trends may be a consequence of individuals ignoring vital information such as the substantial nutrient content as well as the overall balance and low energy density to nutrient density ratio of the potato in addition to other beneficial components.

Compounding this, research has also indicated that the GI of potatoes is high relative to other starches, in spite of recent evidence suggesting a high variability in these measurements or little consideration taken for the preparation method of the potato (potato chips vs. baked potato, for example). Additionally, potatoes are commonly consumed with other foods which in turn often significantly lower the GI of the meal when compared to consumption of the potato alone. For example, Estima potatoes ingested with 62 g of cheddar cheese reduced the GI from 93 to 39 and mashed potatoes served with oil, chicken breast and salad (representing a meal) reduced the GI of the potato from 108 to 54. The GI is based on the consumption of a fixed amount of available carbohydrate, which may not be representative of the glycaemic effect of the amount of carbohydrate usually consumed in a serving of a food within a meal, such as the case with potatoes.

We have extensive experience in conducting experimental studies especially with children. Previously in our laboratory, we investigated and published numerous studies focused on assessing food intake (FI) regulation and appetite in children aged 9 to 13 years.

Thus, the purpose of the current study is to determine effects of commonly consumed carbohydrate sources such as potatoes, pasta and rice along with a fixed portion of meat on blood glucose, satiety and insulin levels among healthy body weight children (aged 11 to 13 years) over a 2 hour period.

ELIGIBILITY:
Inclusion Criteria:

* boys and girls
* age 11 to 13 years old
* healthy
* BMI-for-age percentile 15% to 85%

Exclusion Criteria:

* taking any medications,
* Parental report of children with major disease,
* behavioral or emotional difficulties,
* children who have a food allergy,
* children follow a therapeutic diet, or do not habitually eat breakfast

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Food Intake | Food intake will be measured at 30 min after ad libitum carbohydrate intake
  Food intake (kCal) will be assessed 30 min after consumption of the ad libitum treatments of either rice, pasta, boiled and mashed potatoes, baked french fries or fried french fries.

SECONDARY OUTCOMES:
blood glucose | blood glucose will be measured at 0, 30, 45, 60, 75, 90 and 120 min - during the 2 hours study period.
  Blood glucose (mmol/L) will be measured using finger prick capillary blood samples
Plasma Insulin hormone | Insulin will be measured at 0, 30, 60 and 120 min - during the 2 hours study period.
  Plasma Insulin hormone will be measured using intra-venous blood sample
Plasma Glucogan like peptide (GLP-1) hormone | GLP-1 will be measured at 0, 30, 60 and 120 min - during the 2 hours study period.
  Plasma GLP-1 hormone will be measured using intra-venous blood sample
Plasma ghrelin hormone | Active ghrelin hormone will be measured at 0, 30, 60 and 120 min - during the 2 hours study period.
  Plasma ghrelin hormone will be measured using intra-venous blood sample
Peptide YY (PYY) hormone | PYY hormone will be measured at 0, 30, 60 and 120 min - during the 2 hours study period.
  Plasma PYY hormone will be measured using intra-venous blood sample
subjective appetite | Subjective appetite will be measured at 0, 30, 45, 60, 75, 90 and 120 min - during the 2 hours study period.
  Subjective appetite will be measured by using visual analouge scales

CONTACTS AND LOCATIONS:
Overall Officials: Harvey G Anderson, PhD, Principal Investigator — University of Toronto, Toronto
Locations (1):
- Department of Nutritional Sciences, FitzGerald Building, Toronto, Ontario, Canada